CLINICAL TRIAL: NCT01265251
Title: Evaluation of a Computerised Neuropsychological Test Battery for Idiopathic Normal Pressure Hydrocephalus (INPH)
Brief Title: Computerized Neuropsychology in Idiopathic Normal Pressure Hydrocephalus (INPH)
Status: Completed | Type: Observational
Sponsor: Umeå University (Other)
Responsible Party: Anders Behrens M.D., Department of Clinical Neuroscience
Other Study IDs: 07-088M
Record Dates: First submitted 2010-12-21; First posted 2010-12-23 (Estimated); Last update posted 2010-12-23 (Estimated); Status verified 2010-12

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Normal Pressure Hydrocephalus; Neuropsychological Test; Assessment of cognitive disorders/dementia; Neuropsychological assessment
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Dementia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Test-retest: Forty-four healthy elderly 60-82 years old
  Interventions: Device: Computerized neuropsychological test
- Validity: Twenty six patients with various diseases and various ages
  Interventions: Device: Computerized neuropsychological test; Other: Conventional neuropsychological test
- Feasibility: Twenty seven patients under the preoperative investigation for INPH
  Interventions: Device: Computerized neuropsychological test

INTERVENTIONS:
Device: Computerized neuropsychological test — Computerized neuropsychological test battery.
Other: Conventional neuropsychological test — Conventional neuropsychological test (paper and pen)
  Groups: Validity

SUMMARY:
A computerised neuropsychological test battery to be used as a standardised tool assessing the cognitive domains affected by idiopathic normal pressure hydrocephalus INPH was developed. The aim of this study is to investigate the reliability, validity and feasibility of the battery.

ELIGIBILITY:
Inclusion Criteria:

* Probable INPH under investigation
* Healthy elderly
* Various diseases

Exclusion Criteria:

* (Healthy elderly) medications affecting nervous system
* (Healthy elderly)heart disease
* (Healthy elderly)diabetes
* (Healthy elderly)disease of the nervous system
* (Healthy elderly)MMSE < 28
* (Healthy elderly)vascular risk factors (Two of: 1 hypertension, 2 smoking or 3 hyperlipidemia)
* (Healthy elderly)serious disease that may shorten life expectancy
* (Various diseases) Affected motor functions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Reliability: Healthy elderly Validity: Various diseases Feasibility: Possible INPH-patients
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2007-08; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Validity | Within 24 h
  Computerized test battery and equivalent standard neuropsychological test battery is given to the same subject. Correlation between paper and pen and equivalent computerized test is calculated as a validity measure.
Reliability | More than 7 days, within 2 months
  The computerized test battery is given to the same subject twice. Correlation between the two tests is calculated as a test-retest reliability measure.
Feasibility | Within 24 h
  Patients under the investigation for INPH are given the computerized test battery. Number of patients who manage to complete the test is the feasibility measure.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Behrens, M.D., M.Sc., Principal Investigator — Department of Clinical Neuroscience
Locations (1):
- Department of Clinical Neuroscience, Umeå, Västerbotten County, Sweden

REFERENCES:
- [Derived] Behrens A, Eklund A, Elgh E, Smith C, Williams MA, Malm J. A computerized neuropsychological test battery designed for idiopathic normal pressure hydrocephalus. Fluids Barriers CNS. 2014 Sep 25;11:22. doi: 10.1186/2045-8118-11-22. eCollection 2014. PMID 25279138